CLINICAL TRIAL: NCT07327281
Title: A Phase Ia Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of TQF3250 Capsules in Healthy Adult Subjects After Single Administration and Escalating Doses
Brief Title: A Clinical Trial Evaluating TQF3250 Capsules in Healthy Adult Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQF3250-Ia-01
Record Dates: First submitted 2025-12-05; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQF3250 placebo (Placebo Comparator): Placebo without drug substance.
  Interventions: Drug: TQF3250 placebo
- TQF3250 capsule (Experimental): Oral administration, the fasting administration group was administered once, and the food-influenced group was administered once per cycle, for a total of two cycles. Each cycle is 10 days.
  Interventions: Drug: TQF3250 capsule

INTERVENTIONS:
Drug: TQF3250 placebo — TQF3250 capsule is a biased GLP-1 (glucagon-like peptide-1) receptor agonist developed by Chia Tai Tianqing Pharmaceutical Group Co., Ltd. By binding to the GLP-1 receptor, it can selectively activate certain signaling pathways of the GLP-1 receptor and reduce activation of other pathways, thereby bringing higher efficacy and lower side effects.
  Arms: TQF3250 placebo
Drug: TQF3250 capsule — TQF3250 capsule is a biased GLP-1 (glucagon-like peptide-1) receptor agonist developed by Chia Tai Tianqing Pharmaceutical Group Co., Ltd. By binding to the GLP-1 receptor, it can selectively activate certain signaling pathways of the GLP-1 receptor and reduce activation of other pathways, thereby bringing higher efficacy and lower side effects.
  Arms: TQF3250 capsule

SUMMARY:
TQF3250 capsule is a biased GLP-1 (glucagon-like peptide-1) receptor agonist developed by Chia Tai Tianqing Pharmaceutical Group Co., Ltd. By binding to the GLP-1 receptor, it can selectively activate certain signaling pathways of the GLP-1 receptor and reduce activation of other pathways, thereby bringing higher efficacy and lower side effects.

ELIGIBILITY:
Inclusion Criteria:

* Chinese subjects aged above 18 years old (including 18 years old) and below 55 years old (including 55 years old);
* Those who voluntarily sign a written informed consent form before the trial, have a full understanding of the trial content, process and possible adverse reactions, can communicate well with the researcher, and understand and comply with the requirements of this study;
* Women of childbearing potential should agree to use effective contraceptive measures during the study and for 6 months after the end of the study;
* Male weight ≥50 kg, female weight ≥45 kg, body mass index (BMI) between 20-40kg/m2 (including both ends of the cutoff);

Exclusion Criteria:

* Pregnant and lactating women.
* Those whose vital signs, physical examination, laboratory examination, 12-lead electrocardiogram, anteroposterior chest X-ray, and abdominal ultrasound results during the screening period are abnormal and have clinical significance.
* Those who have had or currently have diseases/abnormalities such as heart, endocrine, metabolism, kidney, liver, gastrointestinal tract, skin, infection, blood, nerve or mental illness, or related chronic diseases, or acute diseases, and the researcher assesses that they are not suitable to participate in the trial:
* Have active tuberculosis during the screening period, or be a close household contact of an untreated active tuberculosis patient.
* Have a history of severe bacterial, fungal or viral infection within 2 months before randomization, requiring hospitalization with intravenous antibiotics or antiviral drug treatment;
* Those who have received major surgical treatment, obvious traumatic injury or major surgery during the expected study treatment within 4 weeks before the first medication (except for the surgery stipulated in the program), or have long-term uncured wounds or fractures;
* Subjects with any bleeding or bleeding events ≥ Common Terminology Criteria (CTC) AE grade 3 within 4 weeks before the first dose;
* Clinically significant infections occur during the screening period, including but not limited to upper respiratory tract infection, lower respiratory tract infection, herpes simplex, herpes zoster, and require antibiotic or antiviral drug treatment.
* Have a history of severe herpes zoster or herpes simplex infection, including but not limited to herpetic encephalitis, disseminated herpes simplex, and generalized herpes zoster.
* Use any systemic cytotoxic or systemic immunosuppressive drugs within 6 months before randomization or within the study period, or use any local cytotoxic or local immunosuppressive drugs within 4 weeks before randomization or within 5 half-lives (whichever is longer) or during the study period.
* Have received any other biological agents on the market or under investigation within 3 months or 5 half-lives (whichever is longer) before randomization.
* Have received a live vaccine within 4 weeks before randomization or plan to receive a live vaccine during the study.
* Those who have undergone surgery within 4 weeks before randomization, or plan to have surgery during the study period.
* Those who lost blood or donated more than 400 mL of blood within 4 weeks before randomization.
* Taking any prescription drugs, non-prescription drugs and herbal medicines within 4 weeks before randomization, except vitamin products.
* Those who have difficulty collecting blood and have a history of fainting from needles or bleeding.
* Are allergic to any known ingredients of TQF3250 capsules, or have any history of severe drug allergy.
* Those with a history of drug abuse or positive urine drug screening.
* Those who smoke more than 5 cigarettes/day or use a considerable amount of nicotine or nicotine-containing products within 3 months before randomization, or who cannot stop using any tobacco products during the trial.
* Those who have been alcoholics for a long time or who drank more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits with an alcohol content of 40% or 150 mL of wine) within 3 months before screening, or who cannot abstain from alcohol during the test, or who have a positive alcohol breath test.
* Those who habitually consume too many caffeinated drinks or foods within 4 weeks before screening. Have consumed grapefruit, bitter orange and the juice of these fruits within 7 days before the first dose, or cannot stop consuming grapefruit, bitter orange and the juice of these fruits during the study;
* Those who have special dietary requirements and cannot accept standard diet;
* There are any other reasonable medical, mental or social reasons that the researcher believes to be unable to participate in this study.
* Those who are unable to comply with the trial plan;
* Those who participated in and used other clinical trial drugs within three months before the first medication;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with incidence and severity of all adverse events (AEs), serious adverse events (SAEs), and treatment-emergent adverse events (TEAEs) | Up to 20 days
  Number of participants with incidence and severity of all adverse events (AEs), serious adverse events (SAEs), and treatment-emergent adverse events (TEAEs).
Number of participants with abnormal clinical laboratory test indicators | Up to 20 days
  Number of participants with abnormal clinical laboratory test indicators.
Changes in body temperature after using TQF3250 capsules | Up to 24 hour
  Evaluate changes in body temperature after using TQF3250 capsules
Tolerance assessment: 12-lead electrocardiogram | Up to 20 days
  Tolerance assessment: 12-lead electrocardiogram
Changes in pulse/heart rate after use of TQF3250 capsules | Up to 24 hour
  Changes in pulse/heart rate after use of TQF3250 capsules
Changes in respiratory rate after using TQF3250 capsules | Up to 24 hour
  Evaluate changes in respiratory rate after using TQF3250 capsules
Changes in blood pressure after using TQF3250 capsules | Up to 24 hour
  To evaluate the changes in blood pressure after using TQF3250 capsules
Changes in blood oxygen saturation after using TQF3250 capsules | Up to 24 hour
  Evaluate changes in blood oxygen saturation after using TQF3250 capsules

SECONDARY OUTCOMES:
Peak drug concentration (Cmax) | Within 20 days after administration
  It refers to the highest blood concentration reached after administration of TQF3250 capsules.
Area under the concentration-time curve from time zero to the last measurable concentration time t (AUC0-t) | Within 20 days after administration
  Area under the concentration-time curve from time zero to the last measurable concentration time t (AUC0-t).
Area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) | Within 20 days after administration
  Area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞).
Peak time (Tmax) | Within 20 days after administration
  It refers to the time it takes for TQF3250 capsules to reach the highest blood concentration after administration.
To evaluate the AUC0-t of TQF3250 capsules and possible metabolites under two administration methods: fasting and postprandial | Up to 20 days
  To evaluate the AUC0-t of TQF3250 capsules and possible metabolites under two administration methods: fasting and postprandial.
To evaluate the AUC0-∞ of TQF3250 capsules and possible metabolites under two administration methods: fasting and postprandial | Up to 20 days
  To evaluate the AUC0-∞ of TQF3250 capsules and possible metabolites under two administration methods: fasting and postprandial.
Evaluate the geometric mean Cmax of TQF3250 capsules and possible metabolites under two administration methods: fasting and postprandial | Up to 20 days
  Evaluate the geometric mean Cmax of TQF3250 capsules and possible metabolites under two administration methods: fasting and postprandial.
Evaluate 90% confidence intervals for TQF3250 capsules and possible metabolites | Up to 20 days
  Evaluate 90% confidence intervals for TQF3250 capsules and possible metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- Drum Tower Hospital Affiliated to Nanjing University School of Medicine, Nanjing, Jiangsu, China